CLINICAL TRIAL: NCT03034291
Title: Controlled Clinical Trial of the Effect of Cocoa Consumption in Patients With Insulin Resistance
Brief Title: Cacao Consumption in Patients With Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cacao IV
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Insulin Resistance
Keywords: Cocoa; obesity; HOMA-IR; BMI; Quality of life
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cacao 70% (Experimental): Consumption for eight weeks of 50 grams of chocolate with 70% cocoa solids equivalent to not less than 430 mg of cocoa polyphenols at each dose.
  Interventions: Dietary Supplement: Cacao 70%
- White chocolate (Placebo Comparator): Consumption for eight weeks of 50 grams of chocolate free of cocoa solids as placebo.
  Interventions: Dietary Supplement: White chocolate

INTERVENTIONS:
Dietary Supplement: Cacao 70% — Consumption for 8 weeks of 50 grams of chocolate per day with 70% cocoa solids.
  Arms: Cacao 70%
Dietary Supplement: White chocolate
  Arms: White chocolate

SUMMARY:
Metabolic syndrome (MS) is a clinical entity that includes several disorders that predispose to imbalance in lipid metabolism: hypertension, insulin resistance, hypertriglyceridemia, obesity and low levels of high density lipoprotein. The SM itself has a great impact on morbidity and mortality and is also related to increased cerebrovascular risk and Diabetes Mellitus 2 (DM2). In Colombia, DM2 is one of the 10 leading causes of illness and death in people over 45 years. It is accepted that insulin resistance is a stage that precedes the onset of DM2, but there are few alternatives to reverse it or prevent its progression to diabetes.

The control of insulin resistance requires increased physical activity, reduced body weight and changes in eating patterns, measures that are not easily adopted in modern Western society.

There is evidence of the effect of chocolate consumption on increasing insulin sensitivity in both hypertensive diabetic patients as well as in normal individuals, apparently because of the ability of cocoa polyphenols to increase the bioavailability of nitric oxide, Formation of reactive species of oxine, optimizing carbohydrate metabolism and modulating insulin-related cellular signaling events.

A prospective, double-blind, placebo-controlled, double-blind clinical trial evaluating the effect of 50 g of chocolate with 70% cocoa solids, which contributes at least 430 mg of polyphenols, is conducted for 8 weeks in The reduction of insulin resistance defined by the reduction of the HOMA-IR index. In addition, there was an increase in arterial reactivity in non-diabetic individuals with central obesity and insulin resistance. Likewise, to infer the effect of this food intervention in the modification of the total cardiometabolic risk of the participants.

DETAILED DESCRIPTION:
RATIONALE Metabolic syndrome (MS) is a clinical entity associated with obesity, insulin resistance (IR), hypertension, hypertriglyceridemia and low HDL. This syndrome promotes the pathophysiological mechanisms of oxidative stress damage, endothelial inflammation, hypercoagulability, atheromatosis and metabolic dysfunction.

In Colombia, morbidity and mortality from chronic diseases related to MS, such as arterial hypertension and type II diabetes mellitus (DM2) represent high costs to the health system due to the direct attention of these diseases as well as their more frequent complications: acute myocardial infarction, cerebrovascular disease, peripheral neuropathy, retinopathy and renal failure. In addition to social costs due to incapacity for work, loss of years of useful life and reduction in the quality of life of patients and their families.

IR biologically precedes the development of DM2 and some authors propose that it is one of the initial manifestations of MS. It is estimated that 25% of individuals with IR will develop DM2 within 3 to 5 years and 50% will retain their IR status. In the global context, it is estimated that in 2010 approximately 344 million people between the ages of 20 and 79, or 7.9% of the population, are estimated to reach 472 million in 2030, that is, 8.4 million of the adult population with the aggravation that the majority will be located in middle to low income countries.

Despite the relevance of IR in the pathophysiology of DM2, since it is its previous stage, there is no public health policies aimed at conducting an active search for the cases and in the event that the diagnosis is made, there are few alternatives to reverse it or prevent its progression to diabetes. Control of IR demands interventions in people's lifestyles such as increased physical activity, reduced body weight and changes in eating patterns, however, despite the effectiveness of these measures, its real impact is low since it involves drastic modifications in the habits of consumer life that characterize modern Western society.

Grassi et al demonstrated in a short-term (15-day) clinical study that the consumption of black chocolate, as opposed to white chocolate, reduces blood glucose and modulates the mean arterial flow in hypertensive patients who have IR.

A parallel, double-blind, prospective, double-blind, placebo-controlled clinical trial evaluating the effect of consumption of 50 g of chocolate with 70% of cocoa solids and providing at least 430 mg of Polyphenols for 8 weeks in the reduction of IR and in the increase of arterial reactivity in non-diabetic individuals with central obesity and IR. Likewise, it is expected to infer the effect of this food intervention in the modification of the total cardiometabolic risk of the participants. This research seeks to corroborate the studies of other groups, to visualize the effects of cocoa over a longer period of time, and in a sample of Colombian population, characterized by a high degree of mestizaje, where the effects may have some nuances different from those Reported with European populations.

THEORETICAL FRAMEWORK

The MS is a clinical entity defined by the WHO in 1998, which includes several disorders that predispose to imbalance in lipid metabolism. To establish the diagnosis, three of five conditions must be met:

1. Elevated serum triglyceride levels (greater than 150mg / dL),
2. Low serum levels of high-density cholesterol (HDL less than 35 mg / dL in men, less than 39 mg / dL in women),
3. Hypertension (SBP greater than 140 mmHg and / or DBP greater than 90 mmHg) or being treated with antihypertensive drugs.
4. High glycemia levels (greater than 100mg / dL) or being treated with hypoglycemic drugs.
5. Obesity (abdominal circumference greater than 90 cm in men, greater than 80 cm in women and / or body mass index greater than 30).

The MS itself has a great impact on morbidity and mortality, and there is evidence of its association with increased cerebrovascular and DM2 risk.

Obesity Obesity is a risk factor for the development of IR, DM2 and MS, and its evaluation is important not only total body fat but also the anatomical distribution of adipose tissue, with particular relevance to visceral deposits for its contribution to resistance to insulin. Epidemiological evidence shows an increase in cardiovascular risk and DM2 in individuals with MS; in addition, mortality from non-cardiovascular causes increases by 2.26-fold in men and 2.78-fold in women not affected by the syndrome, regardless of age, body mass index (BMI), cholesterol levels and smoking.

Studies related to obesity and chronic diseases recommend the use of abdominal circumference as an indicator of central obesity even in people with normal body mass index. Appropriate cutoffs are proposed based on studies on the variability in the risk of chronic diseases in adults by ethnic group. For Colombia, the WHO recommendations were adopted, according to which abdominal perimeters greater than 90 cm and 80 cm in women are compatible with central obesity.

Chocolate and IR Several studies indicate that regular consumption of fruits and vegetables as well as red wine, tea and chocolate may reduce the risk of cardiovascular diseases due to the flavonoids present in these foods. Cacao (Theobroma cacao) is a food that originates in the Americas, containing 6 to 8% of polyphenols, including flavonoids in their monomeric forms: catechin and epicatechin, and their oligomeric forms: procyanidins.

There is epidemiological evidence of the protective factor conferring cocoa consumption on the Kuna indigenous community, in the development of atherosclerotic disease, arterial hypertension and type 2 diabetes mellitus. Grassi and colleagues have demonstrated the effect of chocolate consumption on increasing sensitivity to insulin in both hypertensive diabetic patients as well as in normal individuals. The mechanisms involved in this process seem to be related to the ability of polyphenols to increase the bioavailability of nitric oxide, reduce the formation of reactive species of the oxide, and also have an effect on the metabolism of carbohydrates and the modulation of the pathways of Signaling related to insulin.

IR is defined as decreased sensitivity or response to the metabolic action of insulin. The concept of IR was first proposed in 1936 to describe diabetic patients who required high doses of insulin.

IR plays an important role in the pathophysiology of DM2 and a strong association with obesity, hypertension, coronary disease, dyslipidemia and metabolic syndrome; therefore, it is very important to have tools to quantify the sensitivity or resistance to insulin in humans so that different aspects of this phenomenon can be studied, such as epidemiology, pathophysiological mechanisms, therapeutic outcomes, natural history, among others.

There are different methods for measuring insulin sensitivity / resistance, one of them being direct (hyperinsulinemic/euglycemic clamping) and the rest calculated from basal insulin and glycaemia measurements. Up to now, the clamping continues as the reference diagnostic method, but indirect methods such as QUICKI and the HOMA have a high correlation with the clamping, but only recently validation was started in epidemiological and clinical studies.

Homeostasis Model Assesment (HOMA) Described since 1985, this model takes into account the interaction between glucose and insulin and predicts the steady state of glucose and insulin concentrations in a wide range of possible combinations of IR and beta cell function pancreas. HOMA assumes a feedback loop between the liver and beta cells, meaning that insulin levels depend on the pancreatic response of beta cells to glucose concentration. Therefore, deficient beta cells reflect a decrease in insulin stimulated by glucose and IR is reflected by a decrease in the suppressive effect of insulin on the hepatic production of glucose. HOMA describes this model of insulin/glucose homeostasis through a series of linear equations. The model predicts, in a fasting state, the constant levels of glucose and insulin for any given combination of beta cell function and insulin sensitivity. In practical terms most studies use HOMA as an index to measure IR and its mathematical formula is expressed as the product of fasting glucose and fasting insulin divided by 22.5 which is a constant of normalization.

Chocolate and cardiometabolic risk The Kuna indigenous community living in the San Blas archipelago in Panama has a low frequency of cerebrocardiovascular disease and DM2. This epidemiological picture is attributed to the habitual consumption of large quantities of cocoa-based beverages and not to protective genetic factors.

Cocoa is a food with a high content of polyphenols and is the one with the highest concentration of flavonoids, which are in monomeric form as catechin and epicatequin and as oligomers are procyanidins. Flavonoids in general and cocoa in particular have the ability to lower blood pressure, increase arterial blood flow, reduce oxidation of low-density lipoprotein, reduce platelet aggregability, and increase insulin sensitivity.

It is postulated that the action of cacao involves several mechanisms, including: 1. Reduction of the inflammatory endothelial response involved in the genesis of the atheromatous plaque, which reduces the expression of adhesion molecules necessary for the migration and activation of macrophages and others Phagocytic cells that are the source of reactive oxygen species as well as inflammatory cytokines necessary to perpetuate endothelial injury. 2. Antioxidant capacity that protects from low density lipoprotein peroxidation. 3. Increased activity of endothelial nitric oxide synthase responsible for the production of nitric oxide necessary to preserve the reactivity of arterial flow. 4. Decrease of platelet agreeability at the expense of lower expression of adhesion molecules. And more recently has been described, increased insulin sensitivity.

Principal objective To estimate the changes in IR index (HOMA-IR) and in the modification of cardio metabolic risk in non-diabetic individuals with IR in a controlled clinical trial, after eight weeks of chocolate consumption with 70% of Cocoa solids.

Secondary Objectives

1. Buy the effect of chocolate consumption with or without cocoa solids for 8 weeks on basal and post glucose load in non-diabetic individuals with IR.
2. Compare baseline insulinemia in non-diabetic subjects with IR after eight weeks of consumption of chocolate with or without cocoa solids.
3. To evaluate the effect of the consumption of chocolate with or without cocoa solids in the modulation of the arterial flow of non-diabetic people with IR.
4. To estimate the effect of chocolate consumption with 70% cocoa solids for eight weeks on the modification of the cardio metabolic risk of non-diabetic individuals with IR.
5. Compare the variation in health-related quality of life among people with IR who receive chocolate with cocoa solids and those who receive chocolate free of cocoa solids at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Abdominal circumference greater than 80 cm in women and greater than 90 cm in men
2. HOMA [basal insulin x basal glycemia] / 22.5 equal to or greater than 2.5
3. Basal glycemia normal or compatible with carbohydrate intolerance (baseline glycemia less than 126 mg / dL).
4. Disposition for the consumption of chocolate.
5. Acceptance and signing of informed consent

Exclusion Criteria:

1. Pregnancy
2. Usual consumption of 50 g or more grams of chocolate three or more times per week
3. Insulin application, consumption of metformin or any other hypoglycemic substance.
4. Surgical history of gastric resection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Changes in the insulin resistance index (HOMA-IR) | Baseline and 8 weeks
  Changes HOMA-IR

SECONDARY OUTCOMES:
Anthropometric measurement 1 | 8 weeks
  Body weight (kilograms)
Anthropometric measurement 2 | 8 weeks
  body mass index
Anthropometric measurement 3 | 8 weeks
  abdominal waist (centimeters)
SF-36 Questionnaire of Quality of life | 8 weeks
  Improvement in the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mónica L Giraldo, PhD, Principal Investigator — Universidad de Antioquia

IPD SHARING:
Plan to Share IPD: No